CLINICAL TRIAL: NCT06050005
Title: Knee Functionality Recovery Indicators in Athletes Submitted to Ligamentoplasty of the Anterior Cruciate Ligament
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Sérgio Miguel Loureiro Nuno, MSc in Physical Therapy and Movement Analysis and PhD student in Health Sciences, Universidade da Coruña
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Universidade da Coruña
Record Dates: First submitted 2023-06-13; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Ligament Injury; Ligament Rupture; Ligament Disorders
Keywords: Ligament injury; Preoperative; Postoperative; Functional tests

STUDY DESIGN:
Intervention Model Description: Experimental: rehabilitation activity All participants will be included in this arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental - rehabilitation activity (Experimental): All participants will be included in this arm.
  Interventions: Diagnostic Test: Diagnostic test through functional tests and comparison of scales applied to participants in the pre-surgical and post-surgical period.

INTERVENTIONS:
Diagnostic Test: Diagnostic test through functional tests and comparison of scales applied to participants in the pre-surgical and post-surgical period. — The protocol is based on the ligamentization stages, since the bibliography relates the ligamentization process with rehabilitation. These stages are necrosis, revascularization, cellular priorities and collagen formation, and different care is required for each stage. Taking these aspects into account, the authors developed recommendations to establish a protocol divided by the evaluation phases of the present work. Users should only move on to the next phase if they achieve the expected results, or that makes the total duration of each protocol vary from user to user. tests and scales will be evaluated before surgery, after 6 weeks of surgery and at the end of treatment.

SUMMARY:
Anterior cruciate ligament (ACL) injuries are recurrent, especially in sports. There is still no consensus on the characterization of functional indicators in this clinical condition, as well as their correlation with measuring instruments and clinical functional tests. It is intended to study the changes in functionality of users undergoing this surgery, aiming with functional assessment scales at different times of recovery. This will allow deciding on more adapted recovery strategies, which can meet the musculoskeletal requirements of the user.

DETAILED DESCRIPTION:
It is proposed to carry by carrying out quasi-experimental, quantitative and analytical studies. The sample will consist of athletes who have started recovering from ACL surgery and who meet the previously established inclusion and exclusion criteria.

The study will use and compare functional tests (Star Excursion Balance Test, Lateral Step Down Test and Weight-Bearing Lunge Test) with measurement instruments: Knee and Osteoarthritis Outcome Score (KOOS), Lyshom Knee Scoring Scale, Lower Extremity Functional Score (LEFS), Return to Sport After Injury Scale (ACL-RSI) and IKDC Subjective Knee Evaluation Form.

The intervention will be performed on individual athletes who have had anterior cruciate ligament injury for the first time or recurrence of this ligament in the same knee or injury in the contralateral knee.

ELIGIBILITY:
Inclusion Criteria:

* Start of physiotherapy in the preoperative context and continuation of recovery up to 2 weeks after surgery; age equal to or greater than 18 years; With or without meniscal injury; Be able to correctly fill in the assessment instruments and complete the Informed Consent Form;

Exclusion Criteria:

* Concomitant bilateral injury/history of surgery or contralateral dysfunction; meniscal suture; cartilaginous injury; injury to the internal lateral ligament, external lateral ligament and posterior cruciate ligament; concomitant intra and extra-articular plastic surgery; individuals with recent heart disease, intermittent claudication, neuropathies and cognitive alterations.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Dynamic balance | 1 day before ACL reconstruction surgery
  Change from baseline in a functional test - Y Balance Test - The test should be performed in the following order: Right Anterior, Left Anterior, Right Posteromedial, Left Posteromedial, Right Posterolateral.
  Left Posterolateral
Dynamic balance | At 6 weeks after ACL reconstruction surgery.
  Change from baseline in a functional test - Y Balance Test
Dynamic balance | At 12 weeks after ACL reconstruction surgery.
  Change from baseline in a functional test - Y Balance Test
Dynamic balance | At 24 weeks after ACL reconstruction surgery.
  Change from baseline in a functional test - Y Balance Test
Dynamic knee stability | At 12 weeks after ACL reconstruction surgery.
  Hop test. In this test, the aim is to jump as far as possible with both legs, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg.
Dynamic knee stability | At 24 weeks after ACL reconstruction surgery.
  Single hop test. In this test, the aim is to jump as far as possible on a single leg, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg. The goal is to have a less than 10% difference in hop distance between the injured limb and uninjured limb.
The International Knee Documentation Committee (IKDC) score | 1 day before ACL reconstruction surgery
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.
The International Knee Documentation Committee (IKDC) score | At 6 weeks after ACL reconstruction surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.
The International Knee Documentation Committee (IKDC) score | At 12 weeks after ACL reconstruction surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.
The International Knee Documentation Committee (IKDC) score | At 24 weeks after ACL reconstruction surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 day before ACL reconstruction surgery
  The dimensions from this scale are divided into 5 items (Symptoms, Pain, Activities of Daily Living, Sports and Leisure Activities and Quality of Life) on a positive orientation scale from 0 (extreme knee problems) to 100 (no knee problems).
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 6 weeks after ACL reconstruction surgery.
  The dimensions from this scale are divided into 5 items (Symptoms, Pain, Activities of Daily Living, Sports and Leisure Activities and Quality of Life) on a positive orientation scale from 0 (extreme knee problems) to 100 (no knee problems).
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 12 weeks after ACL reconstruction surgery.
  The dimensions from this scale are divided into 5 items (Symptoms, Pain, Activities of Daily Living, Sports and Leisure Activities and Quality of Life) on a positive orientation scale from 0 (extreme knee problems) to 100 (no knee problems).
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 24 weeks after ACL reconstruction surgery.
  The dimensions from this scale are divided into 5 items (Symptoms, Pain, Activities of Daily Living, Sports and Leisure Activities and Quality of Life) on a positive orientation scale from 0 (extreme knee problems) to 100 (no knee problems).
Lysholm Rating Scale | 1 day before ACL reconstruction surgery
  This scale consists of eight items. It is scored on a scale of 0 to 100 with higher scores indicating fewer symptoms and higher levels of functioning.
Lysholm Rating Scale | At 6 weeks after ACL reconstruction surgery.
  This scale consists of eight items. It is scored on a scale of 0 to 100 with higher scores indicating fewer symptoms and higher levels of functioning.
Lysholm Rating Scale | At 12 weeks after ACL reconstruction surgery.
  This scale consists of eight items. It is scored on a scale of 0 to 100 with higher scores indicating fewer symptoms and higher levels of functioning.
Lysholm Rating Scale | At 24 weeks after ACL reconstruction surgery.
  This scale consists of eight items. It is scored on a scale of 0 to 100 with higher scores indicating fewer symptoms and higher levels of functioning.
Lower Extremity Functional Scale (LEFS) | 1 day before ACL reconstruction surgery
  This measurement instrument consists of 20 items, each of which is scored on a scale five points, from zero to four. The total LEFS score, with a minimum value of zero - low functional level - and maximum of 80 - high functional level, which can be exposed in percentage terms.
Lower Extremity Functional Scale (LEFS) | At 6 weeks after ACL reconstruction surgery.
  This measurement instrument consists of 20 items, each of which is scored on a scale five points, from zero to four. The total LEFS score, with a minimum value of zero - low functional level - and maximum of 80 - high functional level, which can be exposed in percentage terms.
Lower Extremity Functional Scale (LEFS) | At 12 weeks after ACL reconstruction surgery.
  This measurement instrument consists of 20 items, each of which is scored on a scale five points, from zero to four. The total LEFS score, with a minimum value of zero - low functional level - and maximum of 80 - high functional level, which can be exposed in percentage terms.
Lower Extremity Functional Scale (LEFS) | At 24 weeks after ACL reconstruction surgery.
  This measurement instrument consists of 20 items, each of which is scored on a scale five points, from zero to four. The total LEFS score, with a minimum value of zero - low functional level - and maximum of 80 - high functional level, which can be exposed in percentage terms.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | 1 day before ACL reconstruction surgery
  It is a specific 12-item questionnaire assessing the psychological impact (emotions, confidence in performance and evaluation of risk) of returning to sport after ACL reconstruction. Scores range from 0 to 100, and high scores were related to a positive psychological response
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | At 6 weeks after ACL reconstruction surgery.
  It is a specific 12-item questionnaire assessing the psychological impact (emotions, confidence in performance and evaluation of risk) of returning to sport after ACL reconstruction. Scores range from 0 to 100, and high scores were related to a positive psychological response
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | At 12 weeks after ACL reconstruction surgery.
  It is a specific 12-item questionnaire assessing the psychological impact (emotions, confidence in performance and evaluation of risk) of returning to sport after ACL reconstruction. Scores range from 0 to 100, and high scores were related to a positive psychological response
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | At 24 weeks after ACL reconstruction surgery.
  It is a specific 12-item questionnaire assessing the psychological impact (emotions, confidence in performance and evaluation of risk) of returning to sport after ACL reconstruction. Scores range from 0 to 100, and high scores were related to a positive psychological response

CONTACTS AND LOCATIONS:
Overall Officials: Daniel López López, PhD, Study Director — Universidade da Coruña
Locations (1):
- Clínica São João de Deus, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No